CLINICAL TRIAL: NCT00721435
Title: Combined Digital X-ray and Ultrasound Technique for Improved Detection and Characterization of Breast Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Paul L. Carson Ph.D, Principal Investigator, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00045519 (2002-0584); R01CA091713 (NIH)
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Breast Cancer; Mass Cystic; Benign Mass
MeSH Terms: conditions — Breast Neoplasms | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3D Tomosynthesis & 3D Ultrasound for breast masses (Experimental): Evaluate breast screening diagnostic device, 3D tomosynthesis. Assess utility of adding 3D ultrasound.
  Interventions: Procedure: 3D Tomosynthesis and ultrasound imaging
- 3D Tomosynthesis/ 3D Ultrasound for healthy subjects (Experimental): Evaluate breast screening diagnostic device, 3D tomosynthesis. Assess utility of adding 3D ultrasound.
  Interventions: Procedure: 3D Tomosynthesis and ultrasound imaging

INTERVENTIONS:
Procedure: 3D Tomosynthesis and ultrasound imaging — 3D tomosynthesis & ultrasound imaging for scanning masses or healthy breast tissue

SUMMARY:
The study will evaluate and refine a breast screening and diagnosis device.

DETAILED DESCRIPTION:
The device produces 3-D mammograms and ultrasound pictures of the breast at the same time and in the same position. This should help make sure that any area on a mammogram can be easily found in the ultrasound when using the new device. The 3-D mammograms should provide better visualization of the suspected lesion and improve diagnostic accuracy.

ELIGIBILITY:
Inclusion Criteria:

* To participate in this research study you must be a female over the age of 25
* Have had a normal mammogram or are scheduled for a breast biopsy
* Have cysts or have been recommended to have a 6 month follow up mammogram after your biopsy.

Exclusion Criteria:

* Male
* Under the age of 25
* Documented breast cancer

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2002-04; Primary Completion 2014-12 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
To have a device that produces 3D/ultrasound imaging of the breast at the same time and in the same position. | To be determined later.

CONTACTS AND LOCATIONS:
Overall Officials: Paul L Carson, PHD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No